CLINICAL TRIAL: NCT05573737
Title: Investigation of the Effect of Umbilical Cord Care Training Given to Primiparous Mothers on Cord Duration: A Randomized Controlled Study
Brief Title: The Effect of Umbilical Cord Care Training on Cord Falling Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Özlem Selime MERTER, ASSISTANT PROFESSOR, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/ 05- 35
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Umbilical Cord Issue; Mothers; Infant Conditions
Keywords: infant; mothers education; umbilical cord
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Receiving Umbilical Cord Training (Experimental): Oral umbilical care training will be given to the primiparous mothers who gave birth on odd days of the week and met the research criteria, and the training brochure will be printed out and given to the mothers. The training will be given face-to-face during the postpartum period when the mother is stabilized. In order to increase the effectiveness of the training, the content of the training will be reinforced by making mutual questions and answers.
  Interventions: Other: education
- Group Without Umbilical Cord Training (No Intervention): The routine operation of the clinic will be carried out without any intervention for primiparous mothers who gave birth on even days of the week and met the research criteria.

INTERVENTIONS:
Other: education — education about ubilical cord care
  Arms: Group Receiving Umbilical Cord Training

SUMMARY:
Under normal conditions, the umbilical cord is removed 5-15 days after birth. It dries up and falls within days. It is extremely important to determine the factors that cause the prolongation of the falling time of the cord, which poses a serious risk for infection. The aim of this study is to determine the effect of umbilical cord care training given to primiparous mothers on the duration of cord fall. It is a randomized controlled type of research. The population of the research will be primiparous mothers who gave birth in the obstetrics clinic of a university hospital. A pilot study will be conducted to determine the number of samples. As a result of the pilot study, power analysis will be performed and the number of samples will be determined. Inclusion criteria of mothers in the study; Data collection tools: "Descriptive Questionnaire" and "Questionnaire for Umbilical Cord Care" will be used to collect research data. Randomization will be done as odd days of the week and even days of the week for sample selection in the study. Primiparous mothers giving birth on odd days of the week will form the group that will receive umbilical cord training, while primiparous mothers giving birth on even days of the week will form the group that does not receive training. The research will be carried out in two stages. In the first stage of the research, after informing the mothers about the study, they will be invited to the research. Written consent will be obtained from mothers who volunteered to participate in the study. Then, the "Descriptive Questionnaire" prepared to describe mothers and babies will be filled. In the second stage of the research: the mothers will be called 15-20 days after the first interview and the "Question Form Regarding Umbilical Cord Care" will be filled.

DETAILED DESCRIPTION:
Under normal conditions, the umbilical cord is removed 5-15 days after birth. It dries up and falls within days. It is extremely important to determine the factors that cause the prolongation of the falling time of the cord, which poses a serious risk for infection. The aim of this study is to determine the effect of umbilical cord care training given to primiparous mothers on the duration of cord fall. It is a randomized controlled type of research. The population of the research will be primiparous mothers who gave birth in the obstetrics clinic of a university hospital.

A pilot study will be conducted to determine the number of samples. As a result of the pilot study, power analysis will be performed and the number of samples will be determined.

Data Collection:

Stage 1: A pilot study will be conducted with 10 mothers in order to evaluate the appropriateness of the forms and scales used before the research.

Stage 2: The purpose of the research and how to record the data will be explained to the mothers. The mothers in the sample group will be informed about the path followed in practice and the research, and their verbal and written consent will be obtained.

Stage 3:The mothers who meet the sample selection criteria will be randomly and equally distributed into 2 groups through a program in the computer environment, and randomization will be provided.(http://www1.assumption.edu/users/avadum/applets/RandAssign/ GroupGen.html) (1st experimental education group, 2nd control group).

Stage 4: Then, the "Descriptive Questionnaire" prepared to describe mothers and babies will be filled. In the second stage of the research: the mothers will be called 15-20 days after the first interview and the "Question Form Regarding Umbilical Cord Care" will be filled. Umbilical care training will be given to primiparous mothers who give birth on odd days of the week and meet the research criteria, and the training brochure will be printed out and given to mothers. The training will be given face-to-face during the postpartum period when the mother is stabilized. In order to increase the effectiveness of the training, the content of the training will be reinforced by making mutual questions and answers.

The control group will be given routine clinic care. Stage 5: The time of fall of the umbilical cord will be recorded in the data collection form.

Stage 6:The analysis and reporting of the obtained data will be done.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria of mothers in the study;

* Knowing the last menstrual period (SAT),
* Gestational week (GH) interval is due (38-42 GH)
* Able to speak and understand Turkish,
* Not having any chronic disease (diabetes, hypertension, hyper/hypotroid etc.),
* Over 18 years old,
* Normal vaginal delivery
* First born

Exclusion Criteria:

Exclusion criteria for newborns;

* Umbilical cord anomaly (long cord, cord entanglement etc.),
* Needing resuscitation or having a fifth-minute APGAR score of less than 7,
* Birth weight below 2500 g,
* Rh, ABO incompatibility
* Newborns whose umbilical cord does not fall on the postpartum 20th day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
QUESTION FORM FOR UMBLIKAL CORD CARE | 1 day
  It was prepared by researchers in line with the literature in order to evaluate the umbilical cord and care of the baby and to investigate the umbilical fall time. Expert opinion will be taken for the suitability of the form. There are no minimum and maximum scores in the prepared form. The questionnaire are:
  1. Has your baby's umbilical cord fallen off?
  2. Did you close the umbilical cord? 3- Did you bathe your baby before the umbilical cord fell off? 4- If you gave your baby a bath, how did you do it? 5- Have you used any product (alcohol, tenderdiode, ointment, powder, etc.) for your baby's belly care? 6- When tying your baby's diaper, did you pay attention to keep the umbilical cord outside? 7- Has the umbilical cord been in contact with urine or stool? 8- What type of diaper do you use for your baby? 9- Have you had any traditional practices regarding your baby's navel care? 10- What is the baby's diet?

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Karakul, Principal Investigator — Tarsus; Duygu Karaarslan, Principal Investigator — Manisa
Locations (2):
- Turkey (Türkiye) (2):
  - Fırat University, Elâzığ
  - Fırat Univesity, Elâzığ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyngdoh, D., Kaur, S., Kumar, P., Gautam, V., & Ghai, S.(2018). Effect of topical application of human breast milk versus 4% chlorhexidine versus dry cord care on bacterial colonization and clinical outcomes of umbilical cord in preterm newborns. Journal of Clinical Neonatology, 7(1), 25.
- [Background] Oladokun, R. E., Orimadegun, A.E., & Olowu, J. A. (2005). Umbilical Cord Separation Time in Healthy Nigerian Newborns Niger. J Paediatr, 32(1), 19-25.
- [Background] Stewart D, Benitz W; COMMITTEE ON FETUS AND NEWBORN. Umbilical Cord Care in the Newborn Infant. Pediatrics. 2016 Sep;138(3):e20162149. doi: 10.1542/peds.2016-2149. PMID 27573092
- [Background] Nosan G, Paro-Panjan D. Umbilical cord care: national survey, literature review and recommendations. J Matern Fetal Neonatal Med. 2017 Jul;30(14):1655-1658. doi: 10.1080/14767058.2016.1220530. Epub 2016 Aug 23. PMID 27492278
- [Background] Gras-Le Guen C, Caille A, Launay E, Boscher C, Godon N, Savagner C, Descombes E, Gremmo-Feger G, Pladys P, Saillant D, Legrand A, Caillon J, Barbarot S, Roze JC, Giraudeau B. Dry Care Versus Antiseptics for Umbilical Cord Care: A Cluster Randomized Trial. Pediatrics. 2017 Jan;139(1):e20161857. doi: 10.1542/peds.2016-1857. PMID 28008096
- [Background] Ceriani Cernadas JM. Umbilical cord clamping in preterm infants. Arch Argent Pediatr. 2021 Aug;119(4):e315-e321. doi: 10.5546/aap.2021.eng.e315. English, Spanish. PMID 34309309
- [Background] Shang Y, Sun Y. Comparison of the effectiveness of different umbilical cord care in infants: A protocol for systematic review and network meta-analysis. Medicine (Baltimore). 2019 Feb;98(6):e14440. doi: 10.1097/MD.0000000000014440. PMID 30732206
- [Background] Uysal G, Sonmez Duzkaya D. Umbilical Cord Care and Infection Rates in Turkey. J Obstet Gynecol Neonatal Nurs. 2017 May-Jun;46(3):e118-e124. doi: 10.1016/j.jogn.2017.01.008. Epub 2017 Mar 29. PMID 28365249
- [Background] Lopez-Medina MD, Lopez-Araque AB, Linares-Abad M, Lopez-Medina IM. Umbilical cord separation time, predictors and healing complications in newborns with dry care. PLoS One. 2020 Jan 10;15(1):e0227209. doi: 10.1371/journal.pone.0227209. eCollection 2020. PMID 31923218
- [Background] Sachdeva A, Gunasekaran V, Malhotra P, Bhurani D, Yadav SP, Radhakrishnan N, Kalra M, Bhat S, Misra R, Jog P; 'Guidelines on Umbilical Cord Blood Banking' Committee of Indian Academy of Pediatrics. Umbilical Cord Blood Banking: Consensus Statement of the Indian Academy of Pediatrics. Indian Pediatr. 2018 Jun 15;55(6):489-494. PMID 29978816
- [Derived] Merter OS, Karakul A, Karaarslan D, Assistant R. The impact of umbilical cord care education given to Primiparous mothers on cord separation time: A randomized controlled study. J Pediatr Nurs. 2023 Jul-Aug;71:e128-e134. doi: 10.1016/j.pedn.2023.05.005. Epub 2023 May 16. PMID 37202253